CLINICAL TRIAL: NCT00044200
Title: Positron Emission Tomography Imaging of Activation-Induced Signal Transduction in Human Brain
Brief Title: Positron Emission Tomography (PET) to Study Brain Signaling
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000057; 00-N-0057
Record Dates: First submitted 2002-08-21; First posted 2002-08-22 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2015-06-12

CONDITIONS: Healthy
Keywords: Phospholipase A2; Arachidonic Acid; Blood Flow; Coupling; Neurotransmission; PET; Signal Transduction; Activation; Brain; [15O]H20

SUMMARY:
This study uses positron emission tomography (PET) to examine brain function and signaling involving phospholipids, and to see how signaling is related to blood flow. Much of the brain is composed of fatty molecules called phospholipids. These molecules are involved in the way brain cells signal each other to direct brain function. Brain disease may change phospholipids and disturb brain structure and signaling. Studies of brain phospholipid composition and metabolism may help clarify how the brain works in healthy people or stops working effectively in disease states.

Healthy volunteers between 18 and 45 years of age may be eligible for this study. Candidates are screened with a medical history, physical examination, and blood and urine tests. Participants undergo magnetic resonance imaging (MRI) and PET scanning as follows:

MRI

MRI uses a magnetic field and radio waves to produce images of body tissues and organs. For this procedure, the subject lies on a table that is moved into a metal cylinder (the scanner) and wears earplugs to muffle loud knocking and thumping sounds that occur during the scanning process. Scanning time varies from 20 minutes to 3 hours, with most scans lasting between 45 and 90 minutes. Subjects may be asked to lie still for up to 30 minutes at a time.

PET

For the PET scan, a catheter (thin plastic tube) is inserted into an artery in the subject's wrist or elbow crease to collect blood samples during the procedure, and a second catheter is placed in a vein in the opposite arm to inject radioactive tracers. The subject lies on the scanner bed, wearing a special facemask and goggles. The mask helps hold the head still during the scans, and the goggles either block all light or administer bright flashing lights. Radioactive water is injected into the vein, followed by a 1-minute PET scan to measure brain blood flow. This is repeated three more times. Then, a radioactive fatty acid is injected into the vein, followed by a 1-hour PET scan to measure brain phospholipid metabolism. This is repeated once. The images of blood flow and phospholipid metabolism in the different regions of the brain under the conditions of darkness and during visual stimulation provide information on how and where the brain responds to visual stimulation. The entire procedure takes about 3 hours.

DETAILED DESCRIPTION:
Objective

The binding of neurotransmitters and certain drugs to neuroreceptors in the brain is considered to modify cognition and behavior by activating certain receptor-coupled effector enzymes and initiating signal transduction cascades. One of these effector enzymes is phospholipase A2 (PLA2), which when activated will release arachidonic acid (AA) from phospholipids and initiate the AA cascade (Fitzpatrick and Soberman, 2001). AA and its eicosanoid metabolites have multiple biological actions. We have developed an imaging method to quantify and localize brain signal transduction involving PLA2 and AA in unanesthetized rats and monkeys, using quantitative autoradiography or positron emission tomography (PET), and radiolabeled AA. The aim of this protocol is to extend this method to humans with PET, when brain imaging AA signaling in two experimental conditions (dark and visual flash stimulation at a frequency of 3 Hz or 8Hz) in the same subject in the same PET session. Radioactive [1-11C]AA will be injected intravenously in each condition, and PET will be used to measure its incorporation coefficient k* in individual brain regions. Animal studies and modeling have shown that the incorporation coefficient is proportion to PLA2 activation and the release of AA from brain phospholipids (Rapoport, 2003). In addition, [15O]H20 will be injected in each condition to measure regional cerebral blood flow (rCBF). Based on our prior studies in human subjects of rCBF during visual activation by flashing lights at different frequencies (Mentis et al., 1997; Mentis et al., 1998; Mentis et al., 1996), we hypothesize that statistically significant increments in rCBF and [11C]AA incorporation into brain will be increased during visual activation compared with the dark (unactivated) condition. These increments should be evident in primary visual cortex, association visual cortex, thalamus, and frontal cortex. If our hypothesis proves correct and our method to measure [11C]AA incorporation both during stimulation and in the dark proves feasible in the same subject in the PET session, we believe that the method could be applied generally in humans to examine brain PLA2-related signal transduction during physiological or pharmacological activation and in healthy aging (Giovacchini et al., In press) and disease, particularly Parkinson and Alzheimer disease (Hayakawa et al., 2001; Nariai et al., 1991).

Study population

We plan to study 30 normal volunteers, each of whom will be subjected two stimulation conditions in the same PET session, visual stimulation at a frequency of 3 or 8 Hz, or a dark condition (0 Hz).

Design

Each PET scan session will last approximately 3 hours. Each subject will receive a total of four [15O]H20 injections to measure regional cerebral blood flow (rCBF), and two [11C]AA infusions to measure incorporation k* for AA during a single PET scan session. He/she will have an arterial catheter and venous line inserted during the entire session, and one transmission scan at the beginning of the session. The order of the scans will be randomized. The order of 4 blood flow scans will be: Rest-Photic Activation-Photic Activation-Rest OR Photic Activation-Rest-Rest-Photic Activation. The order of two [C11]AA scans will be Rest-Photic Stimulation Or Photic Stimulation-Rest.

Stimulation will be conducted via LED goggles at a flash frequency of 3 Hz and 8 Hz, evenly divided among the 30 subjects, and at 0 Hz (dark condition). Statistical parametric mapping and other statistical procedures will be used to identify brain regions in which k* for AA and/or rCBF is elevated at 3 Hz compared with the dark condition; at 8 Hz compared with the dark condition; and at 8 Hz compared with 3 Hz condition.

ELIGIBILITY:
* INCLUSION CRITERIA:

All subjects must have normal values on screening measures to be in the study.

Age between 18 and 45 years.

EXCLUSION CRITERIA:

Past or current medical condition that would interfere with brain function- history of alcoholism; psychiatric or neurological illness; head trauma with loss of consciousness; history of exposure to central nervous system toxin; history of central nervous system infection; metabolic, endocrine, connective tissue disease; hypertension or other cardiovascular disorder; abnormal renal, liver or pulmonary function; blood or coagulation disease; malignancy; psychopharmacological treatment; neurodegenerative or neurodevelopmental disorder; stroke; epilepsy; sensitivity to flashing lights. Subjects requiring regular medication.

Subjects demonstrated by drug screening to have taken controlled substance.

For female subjects, pregnancy or current breast-feeding (nursing).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2000-01-10; Study Completion 2015-06-12

CONTACTS AND LOCATIONS:
Overall Officials: Stanley I Rapoport, M.D., Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Arai T, Wakabayashi S, Channing MA, Dunn BB, Der MG, Bell JM, Herscovitch P, Eckelman WC, Rapoport SI, Chang MC. Incorporation of [1-carbon-11]palmitate in monkey brain using PET. J Nucl Med. 1995 Dec;36(12):2261-7. PMID 8523117
- [Background] Axelrod J. Phospholipase A2 and G proteins. Trends Neurosci. 1995 Feb;18(2):64-5. doi: 10.1016/0166-2236(95)93873-v. No abstract available. PMID 7537411
- [Background] Axelrod J. Receptor-mediated activation of phospholipase A2 and arachidonic acid release in signal transduction. Biochem Soc Trans. 1990 Aug;18(4):503-7. doi: 10.1042/bst0180503. No abstract available. PMID 2177403